CLINICAL TRIAL: NCT03291782
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, and Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics; Including an Open-label Cohort to Determine the Effect of Food on the Pharmacokinetics of D-0120-NA Tablet in Healthy Volunteers in the United States
Brief Title: D-0120 Safety and PK/PD, Food Effect Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IBIO-201
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- D-0120 Dose 1 (Experimental): D-0120 Dose 1 Patients will get D-0120 single agent or placebo of matching size during dose escalation
  Interventions: Drug: D-0120
- D-0120 Dose 2 (Experimental): D-0120 Dose 2 Patients will get D-0120 single agent or placebo of matching size during dose escalation
  Interventions: Drug: D-0120
- D-0120 Dose 3 (Experimental): D-0120 Dose 3 Patients will get D-0120 single agent or placebo of matching size during dose escalation
  Interventions: Drug: D-0120
- D-0120 Dose 4 (Experimental): D-0120 Dose 4 Patients will get D-0120 single agent or placebo of matching size during dose escalation
  Interventions: Drug: D-0120
- D-0120 Dose 5 (Experimental): D-0120 Dose 5 Patients will get D-0120 single agent once in the fasted state and once in the fed state.
  Interventions: Drug: D-0120

INTERVENTIONS:
Drug: D-0120 — oral, single dose

SUMMARY:
This initial clinical study in the US will be a randomized, double-blind, placebo-controlled, single-dose, dose-escalation, and sequential cohort study to evaluate the safety, tolerability, PK and PD of D-0120-NA in fasting, healthy volunteers (HVs).

In food effect cohort, subjects will each receive 2 doses of D-0120-NA in an open-label manner; once in the fasted state and once in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be medically documented as healthy and acceptable at physical examination.
* Subjects serum uric acid level at screening ≥ 4.5 mg/dL.
* Subjects must have a BMI between 18.0 and 30.0 kg/m2 and a body weight of 50 kg or higher
* Subjects must have all laboratory parameters within the normal range or considered not clinically significant by the principal investigator.
* Subjects must have a normal urinalysis, eGFR, ECG or results considered not clinically significant by the principal investigator.
* Subjects are able to understand the study procedures and risks involved and must provide signed informed consent to participate in the study.

Exclusion Criteria:

* Any history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders.
* Any history or suspicion of kidney stones.
* Positive for HIV, Hepatitis B, and/or Hepatitis C.
* Subjects who have used prescription drugs, over-the-counter drugs, or herbal remedies within 14 days before Day 1 of study medication dosing.
* Undergone major surgery within 3 months prior to Day 1.
* Women who are pregnant or breastfeeding.
* Subjects who received any investigational test article within 5 half-lives or 30 days prior to Day 1 study medication dosing.
* Subjects who consumed Seville oranges- or grapefruit-containing foods or beverages within 7 days before Day 1 and during the entire study duration.
* Subjects with any condition that, in the judgment of the investigator, would place him/her at undue risk, or potentially compromise the results or interpretation of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 weeks
  Adverse Events and changes of Laboratory, Electrocardiogram, and Vital Signs

SECONDARY OUTCOMES:
Pharmacokinetic: area under the plasma concentration versus time curve (AUC) | Day-1 through 3
  AUC: area under the plasma concentration versus time curve for D-0120
Pharmacokinetic: maximum plasma drug concentration (Cmax) | Day-1 through 3
  Cmax: maximum plasma drug concentration of D-0120
Pharmacokinetic: Time to reach the Cmax (Tmax) | Day-1 through 3
  Tmax: Time to reach the Cmax of D-0120
Pharmacokinetic: Apparent terminal half-life (t1/2) | Day-1 through 3
  t1/2: apparent terminal half-life of D-0120
Pharmacokinetic: Apparent oral clearance (CL/F) | Day-1 through 3
  CL/F: Apparent oral clearance of D-0120
Pharmacokinetic: Apparent volume of distribution (Vz/F) | Day-1 through 3
  Vz/F: Apparent volume of distribution of D-0120
PD profile of D-0120 from plasma and urine | Day-1 through 3
  Profile in terms of Serum uric acid and creatinine; Urine uric acid and creatinine. These parameters will be combined to report fractional excretion of uric acid (FEUa %)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Coleman, MD, Principal Investigator — Covance
Locations (1):
- Covance Daytona Beach Clinical Research Unit, Daytona Beach, Florida, United States